CLINICAL TRIAL: NCT01017263
Title: Vyvanse and Glucose Intolerance in Children With ADHD and Obesity
Brief Title: Vyvanse and Glucose Intolerance in Children With Attention Deficit Hyperactivity Disorder (ADHD) and Obesity
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due very high screen fail rate, pre study feasibility not consistent with screened population.
Sponsor: Duke University (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00019063
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2013-09

CONDITIONS: Attention Deficit Hyperactivity Disorder; Glucose Intolerance; Obesity
Keywords: ADHD; Glucose Intolerance; Obesity; Vyvanse
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Glucose Intolerance; Obesity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label Vyvanse (Active Comparator): Eligible subjects will be dispensed open label LDX (VyvanseTM). All subjects will start at 20 mg once a day dose and will be titrated up weekly by 10 mg increments up to a maximum dose of 70 mg. If a subject experiences intolerable side effects at a particular dose, a step down to the next tolerated level is allowed.
  Interventions: Drug: Lis-dexamphetamine

INTERVENTIONS:
Drug: Lis-dexamphetamine — Eligible subjects will be dispensed open label LDX (VyvanseTM). All subjects will start at 20 mg once a day dose and will be titrated up weekly by 10 mg increments up to a maximum dose of 70 mg. If a subject experiences intolerable side effects at a particular dose, a step down to the next tolerated level is allowed.
  Other Names: Vyvanse, LDX

SUMMARY:
The purpose of this study to assess the effects of chronic administration of Vyvanse (lis-dexamphetamine) on glucose metabolism in a sample of children and adolescents with Attention Deficit Hyperactivity Disorder (ADHD) who also have glucose intolerance and are obese.

ELIGIBILITY:
Inclusion Criteria:

* male or female, ages between 8 and 17
* Body Mass Index > 30
* fasting blood sugar between 90-100 mg/dl
* 2 hour post prandial >140 <180 mg/dl
* meets criteria for a diagnosis of ADHD, any subtype

Exclusion Criteria:

* known cardiovascular disease or diabetes
* structural cardiac abnormalities, abnormal ECGs, family history of sudden death
* positive urine drug screen
* fasting blood sugar level > 126 mg/dl
* HbA1c > 6.5 %
* Weight > 300 lbs

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott H Kollins, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Child and Family Study Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants are pre-screened at the Duke Obesity Clinic. Eligible participants then come to the Duke ADHD Clinic for their first study visit.
Pre-assignment Details: At the screening visit, psychiatric evaluation and fasting labs were obtained to determine eligibility. Of the 14 subjects only 2 qualified and received study drug. Reasons for screen fails: 8-did not meet lab parameters for glucose intolerance, 1-elevated BP, 1- elevated TSH, 1- doing well with current ADHD treatment, 1- diagnosed with depression.
Groups:
- Open Label Vyvanse: Eligible subjects will be dispensed open label LDX (Vyvanse). All subjects will start at 20 mg once a day dose and will be titrated up weekly by 10 mg increments up to a maximum dose of 70 mg. If a subject experiences intolerable side effects at a particular dose, a step down to the next tolerated level is allowed.
Period: Overall Study
Arm/Group | Open Label Vyvanse
Started | 14
Completed | 2 (A total of 14 participants screened: 2 qualified and received drug the remaining 12 failed screen)
Not Completed | 12
Not completed — not eligible | 12

BASELINE CHARACTERISTICS:
Groups:
- Open Label Vyvanse: All subjects receive Vyvanse.
Arm/Group | Open Label Vyvanse
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.92 (2.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Pre and Post Study Fasting Blood Sugar and Two Hour Post Prandial.
Description: The study was terminated due to lack of enrollment therefore outcome measures were not assessed. If completed, the expected outcomes would have shown an improvement of the subject's fasting and 2 hour post prandial glucose values, insulin levels and HbA1c. However, all of the subjects recruited did not have abnormal values to start with. The two subjects who were enrolled were the younger kids to which the entry lab criteria do not apply.
Time Frame: Baseline to end of study
Population: Study terminated early - no analysis performed on the single subject with data.
Groups:
- Vyvanse Open Label: Eligible subjects were dispensed open label LDX (VyvanseTM). All subjects started at 20 mg once a day dose and were titrated up weekly by 10 mg increments up to a maximum dose of 70 mg. If a subject experiences intolerable side effects at a particular dose, a step down to the next tolerated level was allowed.
Arm/Group | Vyvanse Open Label
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Open Label Vyvanse
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
Study was terminated due to the high number of failures of lab criteria for glucose intolerance which is one of the entry criterion. No data were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes